CLINICAL TRIAL: NCT01870934
Title: A Feasibility Study on the Development of 3D Optic Ulcer Camera
Brief Title: 3D Camera - Telemedical Foot Ulcer Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Johnny Froekjaer, Research responsible Chief Surgeon, Odense University Hospital
Other Study IDs: OUH3D01; 12-08-00621 (Other: CIV-ID)
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Diabetes Mellitus; Foot Ulcers
Keywords: Telemedicine; Diabetes; Foot Ulcers
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Telemedicine, Diabetes, foot ulcer
  Interventions: Device: Camera

INTERVENTIONS:
Device: Camera — No real intervention, but a comparison of different methods including the new medical device 3D camera.

SUMMARY:
Diabetic foot ulcers are deep wounds that occur as a result of nerve damage in the feet (peripheral neuropathy). Amputation is a common consequence of diabetic foot ulcers; approximately 85% of all diabetes-related amputations are caused by foot ulcers. The ulcer treatment is extensive, resource demanding and highly specialized and necessitates involvement of patient, hospital and local in-home care personnel.

The 3D photo optic camera project aims at a much more efficient and precise method for diagnosis and treatment of foot ulcers. The Department of Endocrinology and the section for LEAN and Innovation at Odense University Hospital has developed a prototype for a 3D camera that takes pictures and measurements of the ulcer that can provide the basis for correct diagnosis and treatment of the ulcer. The camera was developed in close cooperation with TECCLUSTER A/S, Svendborg Municipality, Team Online and ComMed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetic foot ulcers, which has been the diagnosis, stratification (eg ischemia, neuropathy, etc.) and treatment according to current guidelines refer "Diabetic Foot Study Group". Age 18-90 years

Exclusion Criteria:

* Superficial wounds (superficial skin defect with loss of substance in 5 x 5 mm)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic foot ulcers patients
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Comparison of 3D image and normal assessment of wounds | outcome measure is assessed in 2013

SECONDARY OUTCOMES:
Comparison of 3D and 2D image assessment of wounds | november 2013

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Schnack Rasmussen, M.D, Principal Investigator — Odense University Hosptial; Knud Yderstræde, MD, Ph.d., Study Chair — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Odense, Denmark